CLINICAL TRIAL: NCT07244224
Title: The Effect of a Psychosocial Adjustment Program on Healthy Lifestyle Behaviors and Sleep Deprivation in Ninth-Grade Boarding Female Students:A Non-Randomized Controlled Study
Brief Title: The Effect of a Psychosocial Adjustment Program on Healthy Lifestyle Behaviors and Sleep Deprivation in Ninth-Grade Boarding Female Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Habibe Arslan, School Health Nurse, MSc Student in Public Health Nursing, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TBAEK-714
Record Dates: First submitted 2025-09-05; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Lifestyle; Sleep Deprivation; Psychosocial Adjustment
Keywords: Healthy lifestyle study; Boarding high school education; Sleep deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled intervention study with a pre-test, post-test, and follow-up design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Adaptation Program (Experimental): In the study, while the intervention group will participate in a five-day psychosocial adjustment program, no intervention will be conducted in the control group.
  Interventions: Behavioral: Implementation of the Psychosocial Adaptation Program
- Control group (No Intervention): No intervention will be administered to the control group.

INTERVENTIONS:
Behavioral: Implementation of the Psychosocial Adaptation Program — It is a five-day psychosocial adjustment program designed for female boarding high school students. It focuses on promoting healthy lifestyle and improving sleep comfort. The program includes group education sessions and activity-based interventions tailored to this age group.
  Arms: Psychosocial Adaptation Program

SUMMARY:
The World Health Organization defines adolescence as the ages between 10 and 19, emphasizing that supporting both the mental and physical health of this age group is crucial for determining the individual's future quality of life. Problems such as stress, anxiety, depression, maladjustment, substance use, and sleep disorders faced by adolescents can negatively affect the development of healthy lifestyle behaviors.

In this context, students living in boarding school settings represent a more vulnerable group in terms of the need for psychosocial support, as they live away from their families. Boarding students experience difficulties in adaptation due to homesickness, lack of social support, academic pressures, and a strictly regulated lifestyle, and this situation directly affects their health behaviors.

In this study, the effectiveness of a psychosocial adjustment program will be evaluated with intervention and control groups formed on a voluntary basis from ninth-grade female boarding students studying at two public boarding science high schools located in Antalya, Türkiye. The intervention group will participate in a psychosocial adjustment program developed by the researcher, consisting of five sessions, while the control group will not receive any intervention. The program includes structured and interactive group activities on themes such as adopting healthy lifestyle habits, stress and anxiety management, social support, sleep hygiene, effective communication, academic adjustment, and emotional relaxation.

The data will be collected in three phases as pre-test, post-test, and follow-up test; the data collection tools will include the Personal Information Form, the Health-Promoting Lifestyle Profile II (HPLP II), and the Sleep Deprivation Scale for Children and Adolescents. The data will be analyzed using the SPSS program, and depending on normal distribution, parametric or non-parametric tests will be applied. The effect of the intervention will be measured with Cohen's d to calculate the effect size. This study holds original value as it develops a school-based intervention model under the leadership of a school health nurse, and it may provide an innovative contribution based on a holistic nursing approach to adolescents by taking its place among the limited psychosocial intervention studies conducted in boarding school settings.

ELIGIBILITY:
Inclusion criteria Being newly enrolled in the ninth grade Residing in the school dormitory as a boarding student Having a parent/guardian signed informed consent form Not having any absences during the research process Exclusion criteria Those who have not given voluntary consent

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The primary reason for including only female students in the study is to ensure access to the sample group and to maintain the homogeneity of the sample. At the school where the study will be conducted, the girls' dormitory is located very close to the school building, allowing some sessions of the psychosocial adjustment program to be conducted regularly and uninterruptedly after school or in the evening. In contrast, the boys' dormitory is situated at a considerable distance from the school, which would create significant limitations in terms of transportation, safety, and time management for ensuring regular participation. Additionally, due to gender-specific psychosocial developmental differences during adolescence, selecting a homogeneous sample will facilitate the adaptation of the intervention program content and allow its effectiveness to be evaluated in a more controlled manner.
Enrollment: 52 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II | Baseline, 4 weeks after baseline, 17 weeks after baseline
  Healthy Lifestyle Behaviors Scale II: The Healthy Lifestyle Behaviors Scale II is used to evaluate individuals' healthy lifestyle behaviors. The scale consists of a total of 52 items and includes six subscales: spiritual growth, health responsibility, physical activity, nutrition, interpersonal relations, and stress management. The overall score of the scale indicates the level of healthy lifestyle behaviors. As the total score increases, it is interpreted that the individual has more healthy lifestyle behaviors.

SECONDARY OUTCOMES:
Sleep Deprivation Scale for Children and Adolescents | Time Frame: Baseline, 4 weeks after baseline, 17 weeks after baseline
  Sleep Deprivation Scale for Children and Adolescents: This scale is used to assess sleep deprivation in participants. Measurements will be taken before and after the intervention. The scale consists of 15 items rated on a Likert-type scale ranging from "strongly agree" to "strongly disagree." Scores on the scale range from 15 to 60. Higher scores indicate worse sleep deprivation.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe ARSLAN, Study Director — Bağlantısız
Locations (1):
- Akdeniz Üniversitesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study was conducted with adolescent participants, and to protect participant confidentiality, IPD (Individual Participant Data) sharing is not planned.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/
- See also: Relevant publications on the study topic from PubMed — https://pubmed.ncbi.nlm.nih.gov/